CLINICAL TRIAL: NCT03672214
Title: Caesarean Delivery With or Without an Indwelling Bladder Catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Aarhus (Other)
Collaborators: Randers Regional Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1-10-72-113-17_2
Record Dates: First submitted 2018-09-13; First posted 2018-09-14 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2018-09

CONDITIONS: Urinary Tract Infections; Cesarean Section; Infection
MeSH Terms: conditions — Urinary Tract Infections; Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Without placement of a catheter (Experimental): No placement of indwelling catheter prior to Caesarean section
  Interventions: Procedure: Without placement of indwelling catheter
- With placement of a catheter (Active Comparator): Placement of indwelling catheter prior to Caesarean section
  Interventions: Procedure: With placement of indwelling catheter

INTERVENTIONS:
Procedure: Without placement of indwelling catheter — No placement of indwelling catheter prior to Caesarean section
  Arms: Without placement of a catheter
Procedure: With placement of indwelling catheter — Placement of indwelling catheter prior to Caesarean section
  Arms: With placement of a catheter

SUMMARY:
The aim of this study is to compare the incidence of catheter associated culture-based urinary tract infection (UTI) after elective CD with or without preoperative placement of a urinary catheter.

DETAILED DESCRIPTION:
Protokol version 2_13092018 Scientific protocol Caesarean delivery with or without an indwelling bladder catheter. A randomised trial.

Background In 2015, approximately 20% of all pregnant women gave birth by caesarean delivery (CD) in Denmark.

Preoperative preparations for CD include the placement of an indwelling urinary catheter. The rationale behind the procedure is to decrease the risk of surgical injury to a distended bladder and to avoid postoperative urinary retention, but the scientific evidence of the benefit to these matters is not compelling(1). On the other hand, the placement of an indwelling urinary catheter poses a considerable risk of urinary tract infection (UTI) (2), besides the costs associated with delayed ambulation, prolonged hospital stay and catheter associated discomfort to the woman (3, 4) A Cochrane review (1) on indwelling bladder catheter versus no catheter inserted at CD, found that indwelling bladder catheterization was associated with longer time to first spontaneous voiding and more pain/discomfort due to catheterization and/or with first voiding. Furthermore, the women with an indwelling catheter had longer time to ambulation and longer hospital stay. None of the included studies (n=3) in the review reported on bladder injury nor the prespecified criteria for diagnosing UTI and thus no result on UTI as a primary outcome could be obtained. In addition, none of the randomized trials on CD with or without an indwelling bladder catheter were carried out in countries with peri-operative procedures and handling of patients similar to those in Europe.

In a prospective clinical study (5), there were no bladder injuries in 344 women undergoing elective CD without a catheter. UTI was significantly more prevalent in the catheterized group (6%) than in the non-catheterized group (0.58%), P<0.05). In retrospective studies on women undergoing CD with an indwelling catheter, the overall prevalence of bladder injuries is found to be around 0.3%(6, 7).

The aim of this study is to compare the incidence of catheter associated culture- based urinary tract infection (UTI) after elective CD with or without preoperative placement of a urinary catheter.

Statistics Sample size: A power calculation was performed based on a 5.7% incidence of UTI in the catheter group and 0.5% in the non-catheter group(4). With an alpha of 0.05 and a power of 80%, a total of 400 women would have to be included to detect a significant difference in the primary outcome.

The association between the placement of an indwelling urinary catheter during caesarean delivery and the outcomes of interest will be explored using an Intention-to-treat (ITT) analysis. The investigators will perform comparative analyses using multivariate logistic regression with calculation of Odds Ratios with 95% confidence intervals with adjustments for significant differences in baseline characteristics. Subgroup analyses will be performed according to the number of previous CDs No interim analysis will be performed. A local trial steering committee will be appointed.

Side effects, risks, and inconveniences for the project participants

Any inconveniences for the women in the study with providing an extra urinary sample for bacterial culture are very small. Women in the indwelling catheter group receive current standard treatment. Women without a catheter may have an increased risk of:

1. Urinary retention; a known side effect to surgical procedures and regional anaesthesia (9, 10). The women without an indwelling catheter might have a slightly increased risk of urinary retention, but with our postoperative surveillance all cases will be detected and treated in both groups of women.
2. Intraoperative bladder injury; the overall risk is very low (0.3%). In women suspected of peri-operative bladder injury, both with or without an indwelling catheter, methylene blue will be installed into the bladder through an indwelling catheter, which will serve to identify the leak. In case of accidental bladder puncture, surgical repair will be performed immediately.

On the other hand, women without a catheter may have a decreased risk of

1. Urinary tract infection
2. Delayed ambulation
3. Prolonged hospitalization

Information from patient records The participants' medical records are accessed for information on the predefined outcomes; urine test results, any voiding difficulties after CD and catheter removal, information on the surgery, time to ambulation, length of hospital stay, any sign or symptoms of an infection or fever during hospital stay and if there has been any contact to our department after discharge.

Legal considerations The project will be reported to the Danish Data Protection Agency through the joint notifications, Region Midtjylland. The information collected from the project participants will be protected according to Danish law (Lov om behandling af personoplysninger and Sundhedsloven).

Basic information (name, contact information, social security number, previous medical and pregnancy history) is provided by the participants upon inclusion.

Financial compensation The project participants will not receive financial compensation for their participation.

Participant information and inclusion Contact to potential participants is established at a joint information meeting for women booked for planned CD, where verbal and written information about the project will be provided, by a project assistant or a midwife from the delivery ward. Both the assistant and midwife are informed and taught personally by the trial doctor. Thus, women will have the opportunity for reflection at least 4 days before making any decision. Furthermore, the women are offered extended verbal information at the delivery ward, where they are welcome to bring an assessor.

In any need of further information, the women will be given contact information on key persons responsible for the project.

All study participants give oral and written consent at the day of the CD, after at least 4 days of consideration in accordance with the Declaration of Helsinki and Central Denmark Research Ethics Committee.

The women are informed that their consent can be withdrawn at any time.

ELIGIBILITY:
Inclusion Criteria:

* Elective caesarean section.

Exclusion Criteria:

1. Antibiotic therapy during the last week before caesarean section
2. ≥ 3 prior CDs.
3. Contractions or rupture of membranes.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 400 (Estimated)
Dates: Start 2019-06-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of urinary tract infection (UTI). | 3 days
  Urine culture (second day post partum) yielding ≥ 10*5 CFU/ml (of one type of bacteria).

SECONDARY OUTCOMES:
The incidence of UTI later than second day postpartum | 30 days
  Treatment for UTI initiated by a general practitioner or hospital
Any need for catheterization due to postoperative urinary retention | 24 hours
  Any need for catheterization due to postoperative urinary retention
Postpartum blood loss >1000 mL. | 4 hours
  Postpartum blood loss >1000 mL.
Time to ambulation | Up until 48 hours
  From time of birth and until standing or walking
Length of hospital stay | Up until 7 days
  From time of birth and until discharge.
Intraoperative laceration of the bladder | 7 days
  Laceration of bladder during surgery
The incidence of preoperative bacteria in urineculture | 1 day
  Positive urine culture preoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Pinar Bor, MD, Ph.D., Study Chair — Aarhus University and the Region Hospital of Randers
Locations (1):
- The Regional Hospital of Randers, Randers, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Abdel-Aleem H, Aboelnasr MF, Jayousi TM, Habib FA. Indwelling bladder catheterisation as part of intraoperative and postoperative care for caesarean section. Cochrane Database Syst Rev. 2014 Apr 11;2014(4):CD010322. doi: 10.1002/14651858.CD010322.pub2. PMID 24729285
- [Background] Weber DJ, Sickbert-Bennett EE, Gould CV, Brown VM, Huslage K, Rutala WA. Incidence of catheter-associated and non-catheter-associated urinary tract infections in a healthcare system. Infect Control Hosp Epidemiol. 2011 Aug;32(8):822-3. doi: 10.1086/661107. No abstract available. PMID 21768769
- [Background] Ghoreishi J. Indwelling urinary catheters in cesarean delivery. Int J Gynaecol Obstet. 2003 Dec;83(3):267-70. doi: 10.1016/s0020-7292(03)00144-9. PMID 14643036
- [Background] Nasr AM, ElBigawy AF, Abdelamid AE, Al-Khulaidi S, Al-Inany HG, Sayed EH. Evaluation of the use vs nonuse of urinary catheterization during cesarean delivery: a prospective, multicenter, randomized controlled trial. J Perinatol. 2009 Jun;29(6):416-21. doi: 10.1038/jp.2009.4. Epub 2009 Feb 12. PMID 19212327
- [Background] Senanayake H. Elective cesarean section without urethral catheterization. J Obstet Gynaecol Res. 2005 Feb;31(1):32-7. doi: 10.1111/j.1447-0756.2005.00237.x. PMID 15669989
- [Background] Oliphant SS, Bochenska K, Tolge ME, Catov JM, Zyczynski HM. Maternal lower urinary tract injury at the time of Cesarean delivery. Int Urogynecol J. 2014 Dec;25(12):1709-14. doi: 10.1007/s00192-014-2446-2. Epub 2014 Jun 26. PMID 24964762
- [Background] Phipps MG, Watabe B, Clemons JL, Weitzen S, Myers DL. Risk factors for bladder injury during cesarean delivery. Obstet Gynecol. 2005 Jan;105(1):156-60. doi: 10.1097/01.AOG.0000149150.93552.78. PMID 15625157
- [Background] Hansen BS, Soreide E, Warland AM, Nilsen OB. Risk factors of post-operative urinary retention in hospitalised patients. Acta Anaesthesiol Scand. 2011 May;55(5):545-8. doi: 10.1111/j.1399-6576.2011.02416.x. Epub 2011 Mar 21. PMID 21418152
- [Background] Mulder FE, Schoffelmeer MA, Hakvoort RA, Limpens J, Mol BW, van der Post JA, Roovers JP. Risk factors for postpartum urinary retention: a systematic review and meta-analysis. BJOG. 2012 Nov;119(12):1440-6. doi: 10.1111/j.1471-0528.2012.03459.x. Epub 2012 Aug 20. PMID 22900796